CLINICAL TRIAL: NCT04057417
Title: If You Build it, Will They Come?... and Live Longer - A Natural Experiment of an Urban Trail Network Expansion and Cardiovascular Disease
Brief Title: An Urban Trail Network and Cardiovascular Disease: A Natural Experiment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Collaborators: Unity Health Toronto (Other); Ontario Agency for Health Protection and Promotion (Other Government); University of Toronto (Other)
Responsible Party: Principal Investigator, Jon McGavock, Associate Professor, University of Manitoba
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS20928
Record Dates: First submitted 2019-01-29; First posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factor; Diabetes Mellitus
Keywords: physical activity; built environment
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Intervention Model Description: Natural Experiment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urban Trail Expansion (Experimental): Neighbourhoods within 400m to 800m of a neely built greenway, defined as a multi-use concrete/asphalt trail that was >4km in length)
  Interventions: Other: Urban Trail
- Control (No Intervention): Neighbourhoods that are located beyond 400 to 800m of a newly built greenway

INTERVENTIONS:
Other: Urban Trail — A newly built urban trail that was part of a large policy/infrastructure investment from the city/province to enhance the built environment for active transport and recreational physical activity in the city of Winnipeg, Manitoba Canada between 2010 and 2012.
  Arms: Urban Trail Expansion

SUMMARY:
Associations between the built environment and health behaviours are robust, however (1) it remains unclear if the behaviours they elicit lead to meaningful improvements in health outcomes, at the population level and (2) little experimental evidence exists supporting these associations. The primary objective of this study is to capitalize on an urban natural experiment to determine if changing the built environment to support physical activity will (1) reduce the burden of CVD within a population and (2) if it's a cost-effective population intervention. An interrupted time series analysis will be performed over a period of 19 years to determine if the expansion of an urban trail network is associated with reductions in major advserse cardiovascular events (MACE) and CVD-related risk factors within a large urban centre in Canada.

DETAILED DESCRIPTION:
Two different time series methods will be used to estimate the effect of an urban trail expansion (i.e. "intervention") that occured in WInnipeg, Manitoba Canada, between 2010 and 2012. The study is designed to determine if a reduction in Major Adverse Cardiovascular Events (MACE) was observed in neighbourhoods that received the intervention relative to trends among the control neighbourhoods that did not receive the intervention. First, a multi-group segmented regression of interrupted time series data will be used to assess the effect of the intervention on CVD incidence, both immediately (change in level) and over time (change in trend) by creating indicator variables . The level will be the base rate of CVD-related end-points at the beginning of the pre-intervention period (2000) and the value immediately following each change point at which successive segments join until 2010. The trend is the rate of change in MACE end-points (in other words, the slope) during a segment. Autoregressive errors will be modeled to account for correlated outcomes. Second, an autoregressive integrated moving average (ARIMA) model will be fitted for the CVD incidence time series by using the standard approach to identification, estimation, and checking. A trend and periodic seasonal terms will be applied to the entire study period (November 2000 to October 2019). A separate ARIMA model will also be built for the pre-intervention period to forecast CVD evolution of the treated neighbourhoods. The number of CVD end-points prevented by the intervention will be estimated by calculating the difference between the predicted number and the observed number of cases. Should there by difficulty fitting an ARIMA model to a relatively small dataset, exponential smoothing models or the Holt Winters Algorithm will be used. Although they require larger sample sizes, they are ideal for this project as (1) they permit a variety of different types of intervention effect to be modeled explicitly, and (2) they are well suited to forecasting future trends.

ELIGIBILITY:
Inclusion Criteria:

* The entire population of Winnipeg

Exclusion Criteria:

* Individuals < 30 years of age and >65 years of age.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2018-01-05 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | 10 years
  Seasonal incident rates of CVD-related mortality, new hospital admissions for cardiac-related events, valvular disease, ischemic heart disease and stroke

SECONDARY OUTCOMES:
Cardiovascular disease-related risk factors | 10 years
  Seasonal incident rates of diabetes, hypertension, dyslipidemia, gestational diabetes

OTHER OUTCOMES:
Trail counts | 12 months
  User counts on the intervention trails

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Research Institute of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
These data are anonymized within a population health and social repository. Data are available via request to the stewards of the repository - Manitoba Centre for Health Policy (MCHP).

REFERENCES:
- [Derived] McGavock J, Hobin E, Prior HJ, Swanson A, Smith BT, Booth GL, Russell K, Rosella L, Isaranuwatchai W, Whitehouse S, Brunton N, Burchill C. Multi-use physical activity trails in an urban setting and cardiovascular disease: a difference-in-differences analysis of a natural experiment in Winnipeg, Manitoba, Canada. Int J Behav Nutr Phys Act. 2022 Mar 28;19(1):34. doi: 10.1186/s12966-022-01279-z. PMID 35346244
- [Derived] Hobin E, Swanson A, Booth G, Russell K, Rosella LC, Smith BT, Manley E, Isaranuwatchai W, Whitehouse S, Brunton N, McGavock J. Physical activity trails in an urban setting and cardiovascular disease morbidity and mortality in Winnipeg, Manitoba, Canada: a study protocol for a natural experiment. BMJ Open. 2020 Feb 18;10(2):e036602. doi: 10.1136/bmjopen-2019-036602. PMID 32075847